CLINICAL TRIAL: NCT03271021
Title: A Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Efficacy and Safety of Topical Administration of FMX101 for 12 Weeks in the Treatment of Moderate-to-Severe Acne Vulgaris (Study FX2017-22)
Brief Title: A Study to Evaluate the Efficacy and Safety of Topical Administration of FMX101 in the Treatment of Moderate-to-Severe Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX2017-22
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Results first posted 2020-02-21 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMX101, 4% minocycline foam (Experimental): FMX101, 4% minocycline foam applied topically once daily for 12 weeks
  Interventions: Drug: FMX101
- Vehicle foam (Placebo Comparator): Vehicle foam applied topically once daily for 12 weeks
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: FMX101 — FMX101, 4% minocycline foam
  Arms: FMX101, 4% minocycline foam
Drug: Vehicle Foam — Vehicle Foam
  Arms: Vehicle foam

SUMMARY:
A Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Efficacy and Safety of Topical Administration of FMX101 for 12 Weeks in the Treatment of Moderate-to-Severe Acne Vulgaris (Study FX2017-22)

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, vehicle-controlled, 2 arm study to evaluate the safety and efficacy over 12 weeks of FMX101 topical foam containing 4% minocycline compared to vehicle in the treatment of subjects with moderate-to-severe facial acne vulgaris. Qualified subjects will be randomized to receive 1 of the following 2 treatments:

* FMX101 4% minocycline foam
* Vehicle foam

ELIGIBILITY:
Inclusion Criteria:

1. Has facial acne vulgaris with:

   1. 20 to 50 inflammatory lesions (papules, pustules, and nodules)
   2. 25 to 100 non-inflammatory lesions (open and closed comedones)
   3. No more than 2 nodules on the face
   4. IGA score of moderate (3) to severe (4)
2. Willing to use only the supplied non-medicated cleanser (Cetaphil Gentle Skin Cleanser) and to refrain from use of any other acne medication, medicated cleanser, excessive sun exposure, and tanning booths for the duration of the study.

Exclusion Criteria:

1. Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne), or any dermatological condition of the face or facial hair (eg, beard, sideburns, mustache) that could interfere with the clinical evaluations.
2. Sunburn on the face.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1488 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (98):
  - Foamix Investigational Site #376, Phoenix, Arizona
  - Foamix Investigational Site #395, Tucson, Arizona
  - Foamix Investigational Site #315, Bryant, Arkansas
  - Foamix Investigational Site #340, Fort Smith, Arkansas
  - Foamix Investigational SIte #377, Little Rock, Arkansas
  - Foamix Investigational Site #366, Encino, California
  - Foamix Investigational Site #403, Los Angeles, California
  - Foamix Investigational Site #303, Murrieta, California
  - Foamix Investigational Site #369, Northridge, California
  - Foamix Investigational Site #387, Palm Springs, California
  - Foamix Investigational Site #393, Pasadena, California
  - Foamix Investigational Site #380, Poway, California
  - Foamix Investigational Site # 328, Sacramento, California
  - Foamix Investigational Site #313, San Diego, California
  - Foamix Investigational Site #336, San Luis Obispo, California
  - Foamix Investigational Site #309, Santa Ana, California
  - Foamix Investigational Site #325, Santa Monica, California
  - Foamix Investigational Site #375, Temecula, California
  - Foamix Investigational Site #381, Aventura, Florida
  - Foamix Investigational SIte #371, Boca Raton, Florida
  - Foamix Investigational Site #311, Boca Raton, Florida
  - Foamix Investigational Site #398, Brandon, Florida
  - Foamix Investigational Site #329, Clearwater, Florida
  - Foamix Investigational Site #378, Davie, Florida
  - Foamix Investigational Site #396, DeLand, Florida
  - Foamix Investigational Site #392, Doral, Florida
  - Foamix Investigational Site #318, Fort Myers, Florida
  - Foamix Investigational Site #401, Hialeah, Florida
  - Foamix Investigational Site #400, Hialeah, Florida
  - Foamix Investigational Site #383, Lake Worth, Florida
  - Foamix Investigational Site #397, Miami, Florida
  - Foamix Investigational Site #370, Miami, Florida
  - Foamix Investigational Site #346, Miami Lakes, Florida
  - Foamix Investigational Site #347, Miami Lakes, Florida
  - Foamix Investigational Site #306, North Miami Beach, Florida
  - Foamix Investigational Site #312, Ormond Beach, Florida
  - Foamix Investigational Site #362, South Miami, Florida
  - Foamix Investigational SIte #382, Tamarac, Florida
  - Foamix Investigational Site #399, Tampa, Florida
  - Foamix Investigational Site #385, Tampa, Florida
  - Foamix Investigational Site #394, Tampa, Florida
  - Foamix Investigational Site #360, West Palm Beach, Florida
  - Foamix Investigational Site #368, Columbus, Georgia
  - Foamix Investigational Site #336, Sandy Springs, Georgia
  - Foamix Investigational Site #384, Nampa, Idaho
  - Foamix Investigational Site #345, Skokie, Illinois
  - Foamix Investigational Site #390, West Dundee, Illinois
  - Foamix Investigational Site #365, Indianapolis, Indiana
  - Foamix Investigational Site #316, New Albany, Indiana
  - Foamix Investigational Site #361, Plainfield, Indiana
  - Foamix Investigational Site #331, South Bend, Indiana
  - Foamix Investigational Site #320, Louisville, Kentucky
  - Foamix Investigational SIte #367, Louisville, Kentucky
  - Foamix Investigational Site #317, New Orleans, Louisiana
  - Foamix Investigational SIte #373, New Orleans, Louisiana
  - Foamix Investigational Site #388, Glenn Dale, Maryland
  - Foamix Investigational Site #304, Beverly, Massachusetts
  - Foamix Investigational Site #314, Brighton, Massachusetts
  - Foamix Investigational Site #334, Watertown, Massachusetts
  - Foamix Investigational Site #322, Saint Joseph, Missouri
  - Foamix Investigational Site #372, St Louis, Missouri
  - Foamix Investigational Site #391, Lincoln, Nebraska
  - Foamix Investigational Site # 327, Omaha, Nebraska
  - Foamix Investigational Site #332, Las Vegas, Nevada
  - Foamix Investigational Site #344, Portsmouth, New Hampshire
  - Foamix Investigational Site #356, Berlin, New Jersey
  - Foamix Investigational Site #337, Verona, New Jersey
  - Foamix Investigational Site #321, Charlotte, New York
  - Foamix Investigational Site #355, New York, New York
  - Foamix Investigational Site #363, New York, New York
  - Foamix Investigational Site #307, Stony Brook, New York
  - Foamix Investigational Site #350, Charlotte, North Carolina
  - Foamix Investigational Site #348, Winston-Salem, North Carolina
  - Foamix Investigational Site #364, Fargo, North Dakota
  - Foamix Investigational Site #310, Bexley, Ohio
  - Foamix Investigational Site #386, Cincinnati, Ohio
  - Foamix Investigational Site #353, Cleveland, Ohio
  - Foamix Investigational Site #330, Dublin, Ohio
  - Foamix Investigational Site #302, Norman, Oklahoma
  - Foamix Investigational Site #335, Exton, Pennsylvania
  - Foamix Investigational Site #349, Hershey, Pennsylvania
  - Foamix Investigational Site #323, Jenkintown, Pennsylvania
  - Foamix Investigational Site #319, Charleston, South Carolina
  - Foamix Investigational Site #305, Mt. Pleasant, South Carolina
  - Foamix Investigational Site #308, Knoxville, Tennessee
  - Foamix Research Site # 301, Arlington, Texas
  - Foamix Investigational Site #374, Arlington, Texas
  - Foamix Investigational SIte #341, Austin, Texas
  - Foamix Investigational Site #351, Austin, Texas
  - Foamix Investigational Site #402, Bryan, Texas
  - Foamix Investigational Site #358, Dallas, Texas
  - Foamix Investigational Site #333, Houston, Texas
  - Foamix Investigational Site #352, Houston, Texas
  - Foamix Investigational Site # 324, Pflugerville, Texas
  - Foamix Investigational SIte #379, Lynchburg, Virginia
  - Foamix Investigational Site #343, Norfolk, Virginia
  - Foamix Investigational Site #389, Seattle, Washington
  - Foamix Investigational Site #359, Tacoma, Washington

REFERENCES:
- See also: Related Info — http://foamix.co.il/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Started | 738 | 750
Completed | 649 | 644
Not Completed | 89 | 106
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 36 | 53
Not completed — Lost to Follow-up | 34 | 39
Not completed — Protocol Violation | 6 | 4
Not completed — Abnormal Lab Results | 1 | 0
Not completed — Miscellaneous | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam | Total
Number analyzed (Participants) | 738 | 750 | 1488
Age, Customized [Count of Participants; unit: Participants]
  9-12 | 42 | 41 | 83
  13-17 | 321 | 309 | 630
  ≥ 18 | 375 | 400 | 775
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 460 | 469 | 929
  Male | 278 | 281 | 559
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 266 | 252 | 518
  Not Hispanic or Latino | 472 | 498 | 970
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 25 | 29 | 54
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 125 | 144 | 269
  White | 571 | 560 | 1131
  More than one race | 14 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Change From Baseline in the Inflammatory Lesion Count at Week 12.
Description: A decrease in the inflammatory lesion count from Baseline to Week 12.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Lesion Count
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 738 | 750
Lesion Count | 16.39 [15.53 to 17.25] | 12.74 [11.88 to 13.61]

2. Primary Outcome: Investigator Global Assessment (IGA) Treatment Success (Dichotomized as Yes/no) at Week 12, Where Success is Defined as an IGA Score of 0 or 1, and at Least a 2-grade Improvement (Decrease) From Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 738 | 750
participants | 199 | 133

3. Secondary Outcome: The Absolute Change From Baseline in the Non-inflammatory Lesion Count at Week 12
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Lesion Count
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 626 | 622
Lesion Count | 18.80 [17.06 to 20.54] | 15.89 [14.14 to 17.65]

4. Secondary Outcome: The Absolute Change From Baseline in the Inflammatory Lesion Count at Week 9
Time Frame: 9 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Lesion Count
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 738 | 750
Lesion Count | 15.59 [14.80 to 16.38] | 11.72 [10.92 to 12.52]

5. Secondary Outcome: The Absolute Change From Baseline in the Inflammatory Lesion Count at the Interim Visit at Week 6
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Lesion Count
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 738 | 750
Lesion Count | 13.09 [12.29 to 13.89] | 9.57 [8.76 to 110.37]

6. Secondary Outcome: IGA Treatment Success (Dichotomized as Yes/no) at Week 6, Where Success is Defined as an IGA Score of 0 or 1, and at Least a 2-grade Improvement (Decrease) From Baseline at the Interim Visit at Week 6
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 738 | 750
participants | 84 | 46

7. Secondary Outcome: IGA Treatment Success (Dichotomized as Yes/no) at Week 9, Where Success is Defined as an IGA Score of 0 or 1, and at Least a 2-grade Improvement (Decrease) From Baseline at the Interim Visit at Week 9
Time Frame: 9 weeks
Measure: Number; unit: participants
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 738 | 750
participants | 137 | 79

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: Number of participants represents the Safety Population.
Arm/Group | FMX101, 4% Minocycline Foam | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/737 | 0/747
Serious Adverse Events (participants affected / at risk) | 1/737 | 4/747
Other Adverse Events (participants affected / at risk) | 0/737 | 0/747
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMX101, 4% Minocycline Foam (N=737) | Vehicle Foam (N=747)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chron's disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03271021/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT03271021/SAP_001.pdf